CLINICAL TRIAL: NCT05028270
Title: Clinical Study of Superselective Ophthalmic Artery Interventional Chemotherapy for Intraocular Retinoblastoma
Brief Title: Treatment of Intraocular Retinoblastoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-21-06
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-06

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma;Intravenous chemotherapy;Eye protection rate
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Balloon technology: The femoral artery is introduced after the patient is fully anesthetized. First, the 5F-VETERBRAL is introduced under the guidance of the guidance. The common carotid artery and internal carotid artery will be received laterally. After whole-body heparinization, micro-catheter and guide wire technology are used. In the figure below, the proximal end of the 4mm super-form occlusion ball is marked far away from the eye, plugged and sealed, and the guide tube is pushed around in the internal carotid artery. When the occlusion is finished, the internal carotid artery and the ophthalmic artery are not accompanied far away, and the plot is good. The guiding catheter drives the injection of drugs, topotecar, and topotecan for 5 minutes (the suction balloon is opened and blocked, and the infusion is continuous) to complete the infusion.
  Interventions: Procedure: Balloon technology;Microcatheter technology
- Microcatheter technology: The tip of the Marathon microcatheter is placed at the opening of the ophthalmic artery. After the contrast agent is confirmed by hand, the chemotherapeutic drugs The femoral artery is introduced after the patient is fully anesthetized. First, the 5F-VETERBRAL is introduced under the guidance of the guidance. Maphalan, carboplatin, and topotecan are injected sequentially for 30 minutes. Make sure that the tip position of the catheter is not maintained during the injection process. verb: move. After the operation is completed, the blocking balloon is pulled out under the guidance of the guide wire, the arterial sheath is removed, and the femoral artery puncture point is pressed to stop bleeding.

INTERVENTIONS:
Procedure: Balloon technology;Microcatheter technology — Describe each group's intervention in sufficient detail, including how and when to give the intervention Suspend or modify the criteria for interventions that have been assigned to the subject (such as changing the dose of the drug due to hazards or subject requirements or improvement/deterioration of the condition, etc.) Strategies to improve the compliance of intervention programs, and other measures to monitor compliance (such as the return of drug tablets, laboratory inspections, etc.) Related care and interventions allowed or prohibited during the trial
  Groups: Balloon technology

SUMMARY:
This study compares the effects of balloon technology and microcatheter technology on the eye protection rate of neuroblastoma

DETAILED DESCRIPTION:
Retinoblastoma is the most common intraocular malignant tumor in childhood, with an incidence of about 1/15,000-20,000, accounting for 4% of all childhood cancers. All patients with bilateral reticuloblastoma and approximately 10%-15% of children with unilateral disease have germline mutations that can be passed on to their offspring.In developed countries, the survival rate is close to 98%. However, due to the limitations of health care in low-income countries, this proportion is much lower, about 40%. Before the 1990s, retinoblastoma was mainly treated with enucleation and external beam radiation therapy (EBRT). However, these methods are associated with many complications, including vision loss and serious side effects. At present, the first-line conservative treatment of retinoblastoma has changed from EBRT and enucleation to Intravenous chemotherapy (IVC) or intra-arterial chemotherapy (IAC), and it has been consolidated through focal treatment. There are two different surgical procedures for intra-arterial chemotherapy, namely balloon technique and microcatheter technique. Investigators observe their effects through a retrospective case-control study.

ELIGIBILITY:
Inclusion Criteria:

1. 1 year old <age ≤ 18 years old;
2. After biopsy, histopathology and immunohistochemistry tests refer to the COG recommended neuroblastoma diagnostic criteria, pathological classification (INPC), and international neuroblastoma staging (INSS)
3. Patients who were diagnosed with RB for the first time or received chemotherapy in our hospital for the first time after diagnosis
4. ECOG scale (ECOG-PS) ≤ 2;

Exclusion Criteria:

1. No antibiotics and no gastrointestinal surgery within 3 months.
2. Patients with autoimmune diseases;
3. Patients with immunodeficiency;
4. Patients who have been treated for relapsed/refractory diseases; relapsed NB is the appearance of new lesions at the primary site or other sites 4 weeks after the multidisciplinary comprehensive treatment reaches CR. Refractory NB is defined as induced by 2 to 4 courses of treatment The post-effect evaluation is progression disease (PD) during chemotherapy;
5. Multiple organ failure;
6. Uncontrolled infection and diarrhea

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children dignosed retinoblastoma
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2022-06-20 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall success rate | 1 year
  To evaluate the 1-year ocular salvage rate in the treatment of retinoblastoma [ Time Frame: 1 year ] 12-month ocular salvage rate: calculate the number and percentage of subjects who reach 12-month ocular salvage rate, and use the exact probability method to estimate 95% CI.
Second tumor rate | 1 year
  To evaluate the 1-year recurrence of the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Min Shi, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine